CLINICAL TRIAL: NCT05975684
Title: A Randomized Controlled Pilot Trial of Baclofen for Children With Rumination Syndrome
Brief Title: Baclofen for Children With Rumination Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Peter Lu, Associate Professor of Clinical Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00002491
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Rumination Syndrome
MeSH Terms: conditions — Rumination Syndrome | interventions — Baclofen

STUDY DESIGN:
Intervention Model Description: Parallel groups of (a) baclofen or (b) placebo control
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized into one of two parallel groups in 1:1 ratio. The specific details of randomization sequence will be managed by investigational pharmacy. The participant, care provider, and research team are blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Baclofen (Active Comparator): Baclofen 0.5 mg/kg/day up to 15 mg/day divided three times a day in liquid formulation for 4 weeks.
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Matching placebo three times a day in liquid formulation for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — 0.5 mg/kg/day up to 15 mg/day divided three times a day for 4 weeks
  Arms: Baclofen
Drug: Placebo — Placebo three times a day for 4 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about baclofen in pediatric patients with rumination syndrome. The main question it aims to answer is whether baclofen is effective in treating children with rumination syndrome. Participants will be asked to take baclofen or placebo for 4 weeks and fill out surveys regarding symptoms.

DETAILED DESCRIPTION:
Rumination syndrome is a functional gastrointestinal disorder characterized by effortless, repetitive regurgitation of recently ingested meal. The objective of this study is to evaluate the efficacy of baclofen, a GABA-b agonist, in children with rumination syndrome. The investigators hypothesize that children with rumination syndrome who are treated with baclofen in addition to standard behavioral treatment will have greater clinical improvement compared to those who receive placebo.

After enrollment into the study, participants will be randomized into one of two parallel groups in a 1:1 ratio: (a) baclofen or (b) placebo control. The research team will be blinded to randomization. Participants will subsequently meet with investigational pharmacist and receive four-week supply of either baclofen 0.5 mg/kg/day up to 15 mg divided three times a day or matching placebo three times a day in liquid formulation. At baseline, the research team will collect information on demographics, medical, and surgical history, relevant diagnostic testing, and relevant past treatments (including working with a psychologist). Patients/families will complete a baseline questionnaire (rumination severity questions, PedsQL, route of nutrition, medications) and then the patient will start taking study drug or placebo in addition to their usual care as determined by the patient's primary gastroenterologist. Participants/families will complete follow-up questionnaires at week 1, week 2, week 4, and then week 8. The questionnaires will be filled out by the patient or guardian electronically via REDCap. The research team will closely monitor for side effects. In addition to asking about any side effects at follow-up timepoints, the research team will also emphasize that families should contact the team using the research team phone number with any instances of suspected side effects even before the next follow-up timepoint. After the 4-week drug or placebo period, participants are free to start or continue baclofen, or use other treatment modalities, as determined by their primary GI team.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-18 years of age who meets Rome IV diagnostic criteria for rumination syndrome and are see at NCH GI clinic

Exclusion Criteria:

* Patients who have contraindications to baclofen due to medical history and/or current medications
* Patients who are non- English speaking
* Patients who are pregnant

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Vomiting once a week or less | The investigators will assess this specific metric at the end of four weeks.
  Percentage of participants in each group who are vomiting once a week or less. This will be evaluated using a rumination severity survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No